CLINICAL TRIAL: NCT02940990
Title: SBRT in Multi-metastatic NSCLC Patients Which Are Pan-negative for Driver Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Director, Department of Radiation Oncology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHLC007
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: NSCLC; SBRT; GM-CSF
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Placebo Comparator): Participants in the Group A will receive 4-6 cycles of standard two-drug chemotherapy. After that, clinical observation or maintenance chemotherapy will be given.
  Interventions: Drug: two-drug chemotherapy containing platinum, including carboplatin/Cisplatin + pemetrexed/docetaxel/paclitaxel/etoposide/gemcitabine/vinorelbine/albumin-bound paclitaxel
- Group B (Experimental): Participants in the Group B will also receive 4-6 cycles of standard two-drug chemotherapy. However, they will receive an additional treatment of SBRT to primary lesions or metastatic lesions combined with GM-CSF.
  Interventions: Radiation: SBRT concurrent with GM-CSF; Drug: two-drug chemotherapy containing platinum, including carboplatin/Cisplatin + pemetrexed/docetaxel/paclitaxel/etoposide/gemcitabine/vinorelbine/albumin-bound paclitaxel

INTERVENTIONS:
Radiation: SBRT concurrent with GM-CSF — SBRT and GM-CSF 125ug/m2 for 14 days
  Arms: Group B
Drug: two-drug chemotherapy containing platinum, including carboplatin/Cisplatin + pemetrexed/docetaxel/paclitaxel/etoposide/gemcitabine/vinorelbine/albumin-bound paclitaxel — two-drug regimen

SUMMARY:
This protocol is a phase II multi-center randomized controlled trial (RCT) evaluating the efficacy of SBRT in multi-metastatic NSCLC patients who are pan-negative for driver mutations.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death. Forty percent of patients are diagnosed as metastatic lung cancer, and about 50% of them are pan-negative for driver mutations. The median overall survival(OS) for these patients is 11 months, and maintenance therapy can only prolong 2 months of OS. The NCCN guidelines recommend 4-6 cycles of chemotherapy with or without maintenance chemotherapy.

Published data showed that radiotherapy modulates tumor phenotypes, enhances antigen presentation and tumor immunogenicity. The regression of out-field lesions was termed as "abscopal effect". The combination of radiotherapy with immunotherapeutic agents may promote the host anti-tumor immune response and increase the rate of abscopal effect.Published data showed that abscopal effect appeared in 20%-30% patients with metastatic malignant tumors who were treated with the combination of SBRT and GM-CSF.

The investigators evaluate the efficacy of the combination of SBRT and GM-CSF in the multi-metastatic NSCLC participants who are pan-negative for driver mutations. Patients enrolled will be randomized into two groups. The control group will receive the standard regimen as NCCN recommends. The experimental group will receive both the standard chemotherapy and the extra SBRT to primary lesions or metastatic lesions combined with GM-CSF. The investigators compare progress free survival(PFS) of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small-cell lung cancer.
* Stage IV according to UICC stage system(version 7,2009).The number of metastatic lesions>5
* Pan-negative for driver mutations including EGFR ALK ROS1 c-MET
* At least Three evaluable lesions among which at least two must be suitable for SBRT.
* ECOG performance status 0-2.
* Expected lifespan ≥3 months.
* No brain metastasis in MRI.
* No liver metastasis in abdominal CT or MRI.
* No malignant pleural effusion or pericardial effusion from chest CT and/or pathology.
* Stable lab values: Hematological:

Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin ≥9 g/dL Renal: Creatinine OR Measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5× the upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels >1.5× institutional ULN Hepatic: Total bilirubin ≤1.5×ULN OR Direct bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN OR ≤5×ULN for patients with liver metastases ,globulin≥20 g/L, albumin≥30 g/L.

- Able to understand and give written informed consent and comply with study procedures.

Exclusion Criteria:

* Any unstable systemic disease, including active infection, uncontrolled high blood pressure, unstable angina, newly observed angina pectoris within the past 3 months, congestive heart failure (New York heart association (NYHA) class II or higher), myocardial infarction onset six months before included into the group, and severe arrhythmia, liver, kidney, or metabolic disease in need of drug therapy.
* Previously diagnosed with immunodeficiency disease.
* Human immunodeficiency virus (HIV) infection.
* Women in pregnancy or lactation .
* Patients with mental illness, considered as "can't fully understand the issues of this research".
* other Cancer history.
* Histologically confirmed small cell carcinoma or other non NSCLC compositions in the cancer tissue.
* Brain metastasis or liver metastasis or malignant pleural effusion or pericardial effusion.
* Allergy of rhGM-CSF and its accessories.
* Contraindications to GM-CSF treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 2 years

SECONDARY OUTCOMES:
Overall Survival （OS） | 2 years
Incidence of treatment-related adverse events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Result] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Result] Stamell EF, Wolchok JD, Gnjatic S, Lee NY, Brownell I. The abscopal effect associated with a systemic anti-melanoma immune response. Int J Radiat Oncol Biol Phys. 2013 Feb 1;85(2):293-5. doi: 10.1016/j.ijrobp.2012.03.017. Epub 2012 May 5. PMID 22560555
- [Result] Daly ME, Monjazeb AM, Kelly K. Clinical Trials Integrating Immunotherapy and Radiation for Non-Small-Cell Lung Cancer. J Thorac Oncol. 2015 Dec;10(12):1685-93. doi: 10.1097/JTO.0000000000000686. PMID 26484629
- [Result] Abuodeh Y, Venkat P, Kim S. Systematic review of case reports on the abscopal effect. Curr Probl Cancer. 2016 Jan-Feb;40(1):25-37. doi: 10.1016/j.currproblcancer.2015.10.001. Epub 2015 Oct 9. PMID 26582738